CLINICAL TRIAL: NCT02881879
Title: An Open, Multicenter Clinical Trial With Subcutaneous Immunotherapy in Depot Presentation in Patients With Allergic Rhinoconjunctivitis Sensitized to House
Brief Title: Clinical Trial With Subcutaneous Immunotherapy in Depot Presentation in Patients With Allergic Rhinoconjunctivitis Sensitized to House Dust Mites
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roxall Medicina España S.A (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIA-HDMD-101
Record Dates: First submitted 2016-07-29; First posted 2016-08-29 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Allergic Rhinoconjunctivitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Allergovac depot with HDM extract (Experimental): Extract of mixture of Dermatophagoides pteronyssinus and Dermatophagoides farinae (50:50) adsorbed onto aluminum hydroxide 0.33%.
  Interventions: Biological: Allergovac depot DPT/DF (50:50)

INTERVENTIONS:
Biological: Allergovac depot DPT/DF (50:50) — Subcutaneous immunotherapy in depot presentation in a rapid dose escalation scheme: 6 weekly dose increasing injections at the initiation phase plus 3 maintenance monthly injections

SUMMARY:
The aim of the study is to evaluate the safety and tolerability of subcutaneous immunotherapy (SCIT) with House Dust Mite (HDM) extract in patients with rhinoconjunctivitis with or without associated mild asthma and sensitized to HDM. In addition,surrogate efficacy parameters will be evaluated: immunoglobulin level changes and skin reactivity.

It will be recruited 50 patients susceptible to receive SCIT with HDM extract along 5 participating spanish sites.

Primary endpoint of the study is to assess the safety and tolerability of subcutaneous immunotherapy in depot presentation and quick pattern in patients with rhinoconjunctivitis with or without mild asthma sensitized to house dust mites

Secondary objective is to evaluate the indirect immunotherapy efficacy through the measurement of immunoglobulin level changes and cutaneous reactivity

DETAILED DESCRIPTION:
The aim of present clinical trial is to go deeper into the safety of the vaccine of mixture of DPT and DF (50:50). Although this is the first clinical trial to date to be performed with this vaccine, there have been two clinical trials with the same formulation and DPT 100% as active ingredient( NºEudraCT: 2009-016277-15 and NºEudraCT: 2011-004583-30). Given that there is a remarkable cross-reactivity between the DPT and DF mites, the results of the two clinical trials conducted to date with subcutaneous depot vaccine with Dermatophagoides pteronyssinus 100% extract mite, are very significant

ELIGIBILITY:
Inclusion Criteria:

1. Patients must sign the informed consent form
2. Patients must be between 18 and 60 years of age
3. Patients with perennial allergic rhinoconjunctivitis against HDM during a minimum of 1 year prior to study participation. Although allergic rhinoconjunctivitis is the pathology under study, the inclusion of patients with mild concomitant asthma is allowed (GINA 2015)
4. Patients who obtained a prick test result ≥ 3 mm diameter to HDM. Positive and negative control of the test should give consistent results
5. Patients with specific immunoglobulin E ≥ class 2 (CAP/PHADIA) to HDM
6. Patients sensitized to HDM with clinically relevant symptoms in which treatment with HDM (50:50) vaccine is indicated
7. Women of childbearing potential must have a negative urine pregnancy test at visit 1
8. Women of childbearing potential must agree to use an appropriate contraception method during the study if they are sexually active

Exclusion Criteria:

1. Patients who received immunotherapy in the previous 5 years for HDM or for any allergen with cross reactivity or patients that are currently receiving immunotherapy for any allergen
2. Patients with severe asthma or forced expiratory volume in 1 second FEV1 < 70% even if the are pharmacologically controlled
3. Polysensitized patients besides other airborne allergens Dermatophagoides pteronyssinus and Dermatophagoides farinae, which according to the investigator may present clinically relevant to those other airborne allergens while participating in this study
4. Patients with: immunological, cardiac, renal or hepatic illnesses or any other medical condition that the investigator deems relevant so as to interfere with the study
5. Patients with a previous history of anaphylaxis
6. Patients with active chronic urticaria
7. Patients with active severe atopic eczema
8. Patients who have participated in another clinical trial within 3 month prior to enrollment
9. Patients under treatment with tricyclic antidepressives, phenothiazines, β- blockers, or Angiotensin Converting Enzyme Inhibitors (ACEI)
10. Female patients who are pregnant or breast-feeding
11. Patient who does not attend the visits
12. Patient's lack of collaboration or refusal to participate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | From date inform consent is signed until the date the treatment is completed, assessed up to 5 months

SECONDARY OUTCOMES:
Immunoglobulin level changes | Prior starting the treatment (baseline) versus one week after the last dose is administered (final visit)
Skin prick test reactivity | Prior starting the treatment (baseline) versus one week after the last dose is administered (final visit)

CONTACTS AND LOCATIONS:
Overall Officials: Araitz Landeta, Study Chair — Roxall Medicina España S.A
Locations (5):
- Spain (5):
  - Hospital Germans Triasl i Pujol, Badalona, Barcelona
  - Hospital de Bellvitge, Barcelona
  - Hospital de Basurto, Bilbao
  - Hospital de Valdecilla, Santander
  - Hospital Universitario de Araba, Vitoria-Gasteiz

IPD SHARING:
Plan to Share IPD: No